CLINICAL TRIAL: NCT02902874
Title: Study of the Biological Mechanisms Associated With the Immunogenicity in Anaplastic Large Cell Lymphoma ( ALCL ) ALK +
Acronym: Immuno ALCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-A01343-54; 2009/1603 (Other: CSET Number)
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: ALCL
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients treated for anaplastic large cell lymphoma ( ALCL ) (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
To study the correlation between the polymorphism of the main immunity genes and progression-free survival in ALCL of the child.

ELIGIBILITY:
Inclusion Criteria:

* Every patients treated according to COPAD-IGR, HM 89,91 and 97 and ALCL99 protocols and included in related studies
* Clinical data registered in SFCE database
* Signed consent form

Exclusion Criteria:

* No ALK expression on tumour
* No consent signed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2010-04-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of single nucleotide polymorphisms in main immunogenicity genes using VERACODE ILLUMINA technology | up to 78 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No